CLINICAL TRIAL: NCT03680196
Title: The Effect of Botulinum Toxin Injection at Hip Adductor Muscles in Patients With Spastic Cerebral Palsy, Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ju Seok Ryu (Other)
Responsible Party: Sponsor-Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1807-478-001
Record Dates: First submitted 2018-09-12; First posted 2018-09-21 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy
Keywords: hip dislocation; GMFCS level 3,4,5
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cerebral palsy patients (Experimental): cerebral palsy patients who have GMFCS level3,4,5 and 2 years old and under 10 years old apply an A injection of medication Botulinum A injection
  Interventions: Drug: medication Botulinum A injection.

INTERVENTIONS:
Drug: medication Botulinum A injection. — In cerebral palsy patients, Botulinum toxin within the allowable dose of 16 U / kg per body weight will injected into both adductor longus, adductor magnus muscle at 3 U / kg, adductor brevis, and gracilis muscle at a dose of 1 U / kg.

SUMMARY:
In children with cerebral palsy, secondary problems lead to hip dislocation. the purpose of this study is to find out the effects of botulinum toxin A on hip joint dislocation in cerebral palsy patients.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of patient group: who has a cerebral palsy and GMFCS level 3,4,5
* Intervention: applied medication Botulinum A injection (meditox 200unit)
* Main outcome measures: The investigators will measure for finding evidence by checking the x-ray photograph, hip adductor and muscles pressure test and electromyography(EMG test) test of hip adductor, abductor and spine muscles.

ELIGIBILITY:
Inclusion Criteria:

* Severe cerebral palsy patients(GMFCS level 3,4,5)
* 2 to 10 years old

Exclusion Criteria:

* Those who disagree with the study.
* other than cerebral palsy.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change from hip adductor and spin muscles electromyography(EMG) test at a month | once at study, when patient enrolled and every once a month for one year
  Use EMG to check the activity of the hip adductor and spine muscles of participants.
  This figures will give investigators a look at the association with a hip dislocation.

SECONDARY OUTCOMES:
Whole spine AP and total Hip AP X-ray photograph | once at study, when patient enrolled and and after six month for one year
  Whole spine and total Hip joint are checked with X-ray photograph. and investigators will check the progress of hip dislocation and spinal scoliosis.
hip adductor muscles pressure meter test | once at study, when patient enrolled and every once a month for one year
  Pressures of hip adductors muscles are measured from pressure meter. and This figures will give investigators a look at the association with a hip dislocation.
Likert scale | once at study, when patient enrolled and every once a month for one year
  Evaluate the satisfaction of botulinum toxin A injection. Likert scale is a response category that indicates the extent to which the question is for or against. Example) Very satisfied - normal - slightly dissatisfied - very dissatisfied
Hip and knee joint Range of motion(ROM) test | once at study, when patient enrolled and every once a month for one year
  Measure the range of motion the knee and hip joints.
CPCHILD sacle | once at study, when patient enrolled and every once a month for one year
  Evaluate the quality of life for patients with cerebral palsy. CPCHILD scale have 6section and each section measures scores by 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea